CLINICAL TRIAL: NCT05317988
Title: Online Training for the Reconstitution of Fosun/BioNTech: a Learning Platform to Determine Readiness for Complex Medication Preparation Procedures
Brief Title: Online Training for the Reconstitution of Fosun/BioNTech
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. Esther Wai Yin Chan, Associate Professor, The University of Hong Kong
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: TDGCOVID-EWC-06-2021
Record Dates: First submitted 2022-04-06; First posted 2022-04-08 (Actual); Last update posted 2023-05-10 (Actual); Status verified 2023-05

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — Control Groups

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Participants receive a step-by-step demonstration video of detailed reconstitution procedures and text-based vaccine product information
  Interventions: Behavioral: Intervention group
- Control group (Placebo Comparator): Participants receive a generic video of similar duration on basic facts of COVID-19 (unrelated to reconstitution procedures) and text-based product information
  Interventions: Behavioral: Control group

INTERVENTIONS:
Behavioral: Intervention group — Participants receive a step-by-step demonstration video of detailed reconstitution procedures and text-based vaccine product information
  Arms: Intervention group
Behavioral: Control group — Participants receive a generic video of similar duration on basic facts of COVID-19 (unrelated to reconstitution procedures) and text-based product information
  Arms: Control group

SUMMARY:
The COVID-19 vaccine by BioNTech requires specific, delicate storage and dilution procedures to be stringently followed for safety and effectiveness. Training should be completed prior to undertaking dilution procedures. Currently, the nursing and pharmacy curricula do not have content on specialized vaccine reconstitution techniques. E-learning has become an essential component of teaching and learning due to COVID. Yet, optimal online learning module development for clinical procedural skill acquisition and appropriate online formative assessment has not been adequately explored. To bridge this training gap for Hong Kong nurses and pharmacists, this project aims to develop a video-based online learning programme, coupled to a randomized controlled study to determine the effectiveness of online vaccine reconstitution training. The module, a supplement to the current teaching curriculum, will train students from both Nursing and Pharmacy disciplines. Outcome measures include formative assessment of student performance, which can be used to inform the design and content of experiential content in healthcare professional curriculums. If this learning platform is shown to be effective, the scope could be extended to other disciplines (not limited to healthcare) where learning complex procedural tasks are necessary for the absence of instructor-led teaching.

ELIGIBILITY:
Inclusion Criteria:

* Students currently enrolled in the Bachelor of Pharmacy and Bachelor of Nursing programmes (Years 1 to 4) at The University of Hong Kong

Exclusion Criteria:

* Students not from the aforementioned programmes and years of study

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 385 (Actual)
Dates: Start 2022-03-28 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Factual knowledge | 1 week
  Students will complete a set of validated multiple-choice questions before and after the training.

SECONDARY OUTCOMES:
Procedural knowledge | 1 week
  Students will complete an interactive psychomotor assessment, where they must sort out the correct sequence of reconstitution procedures using a drag-and-drop interface with instant formative feedback
Self-efficacy | 1 week
  Students will rate their confidence on carrying out the reconstitution procedures in practice before and after the training based on a 10-point Likert scale

CONTACTS AND LOCATIONS:
Locations (1):
- Centre of Safe Medication Practice and Research, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No